CLINICAL TRIAL: NCT01082744
Title: Thoracic Paravertebral Block: a Comparative Study of Ropivacaine With Ropivacaine and Sufentanil for Treating Pain After Video-assisted Thoracic Surgery.
Brief Title: Thoracic Paravertebral Block for Postoperative Analgesia After Video-assisted Thoracic Surgery.
Acronym: PARAVI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009.558; 2009-014832-38 (EudraCT Number)
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Pain, Postoperative
Keywords: Paravertebral Block; Regional Anesthesia; Anesthetics Local; Ropivacaine; Sufentanil; Pain Postoperative; Chronic Pain; Thoracic Surgery Video-Assisted.
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain | interventions — Ropivacaine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous paravertebral block with ropivacaine (Active Comparator)
  Interventions: Drug: Ropivacaine
- Continuous paravertebral block with ropivacaine and sufentanil (Experimental)
  Interventions: Drug: Ropivacaine + Sufentanil

INTERVENTIONS:
Drug: Ropivacaine + Sufentanil — Sufentanil at 0.25 µg/ml added to ropivacaine at 2 mg/ml at a perfusion rate of 0.15 ml/kg/h for continuous paravertebral block over 48 hours
  Arms: Continuous paravertebral block with ropivacaine and sufentanil
Drug: Ropivacaine — Ropivacaine at 2 mg/ml at a perfusion rate of 0.15 ml/kg/h for continuous paravertebral block over 48 hours
  Arms: Continuous paravertebral block with ropivacaine

SUMMARY:
The use of paravertebral catheters is a recommended technique to achieve postoperative analgesia after thoracic surgery. To date there is no consensus on which drug regime (local anesthetics with or without opioid) is best. The aim of this prospective clinical trial is to determine wether the use of ropivacaine and sufentanil injected through a thoracic paravertebral catheter results in decreased acute postoperative pain compared with plain ropivacaine in patients after thoracoscopic lung surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for planned video-assisted thoracic surgery
* Patient that consent to participate
* Planned placement of paravertebral catheter
* Patient having a medical insurance

Exclusion Criteria:

* Patient less than 18 years
* Refusal to participate
* Known pregnancy
* Known allergies to local anesthetics, sufentanil and /or to iodinated contrast material
* Intolerance to sufentanil and/or morphine
* Chronic consumption of opiates
* Preoperative chronic pain syndrome
* Patient having a contraindication to placement of paravertebrtal catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-03; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
morphine consumption during the first 48 hours | 48 hours

SECONDARY OUTCOMES:
Acute pain | 48 hours
  using the Visual Analogue Scale (VAS) score
Biological measurements | 48 hours
  Oxygen saturation, level of sedation, respiratory rate, nausea, vomiting, itching, urine retention, blood pressure, heart rate
Patient satisfaction | 48 hours
Chronic pain | 3 and 6 monthes
  assessed with the Saint-Antoine Pain Questionnaire (French version of the Mac Gill Pain Questionnaire) and the DN4 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Christian BAUER, MD, Principal Investigator — Hospices Civils de Lyon, Hopital Louis Pradel
Locations (1):
- Hospices Civils de Lyon, Hopital Louis Pradel, Department of Anesthesiology, Bron, France

REFERENCES:
- [Result] Bauer C, Pavlakovic I, Mercier C, Maury JM, Koffel C, Roy P, Fellahi JL. Adding sufentanil to ropivacaine in continuous thoracic paravertebral block fails to improve analgesia after video-assisted thoracic surgery: A randomised controlled trial. Eur J Anaesthesiol. 2018 Oct;35(10):766-773. doi: 10.1097/EJA.0000000000000777. PMID 29373333